CLINICAL TRIAL: NCT01409356
Title: Effects of Weight Loss on Portal Pressure in Patients With Compensated Cirrhosis and Overweight/Obesity
Brief Title: Effects of Weight Loss on Portal Pressure in Patients With Overweight/Obesity and Cirrhosis
Acronym: SPORTDIET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Principal Investigator, Jaime Bosch, Prof., Hospital Clinic of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPORTDIET
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Compensated Cirrhosis; Obesity
Keywords: Obesity; Portal hypertension; Cirrhosis; Diet; Exercise
MeSH Terms: conditions — Obesity; Hypertension, Portal; Fibrosis; Motor Activity | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diet+Exercise (Experimental): Program of weight loss through diet+exercise (=intervention)
  Interventions: Behavioral: Diet + exercise

INTERVENTIONS:
Behavioral: Diet + exercise — Program of dietary counselling by dietists, who will periodically follow-up the patient to achieve weight loss; moreover a fitness professional will instruct and train the patients twice a week to enhance their physical activity. A step counter will be also given to all participants and daily step count will be recorded. The duration of diet+exercise is 4 months from baseline HVPG measurement.

SUMMARY:
Overweight/obesity is increasing both in the general population and in patients with cirrhosis. In compensated patients with cirrhosis increased BMI is a risk factor for clinical decompensation independent of liver function and portal pressure. Nonetheless, patients with cirrhosis and obesity show a progressive increase in portal pressure, which might explain their increased risk of complications. Since obesity is a potentially modifiable risk factor, we designed this proof-of-concept study to assess the effects of weight loss (obtained by 4 months of diet and exercise) on portal pressure in patients with compensated cirrhosis and overweight/obesity.

DETAILED DESCRIPTION:
Overweight and obesity markedly increase the risk of appearance and progression of most chronic diseases, including chronic liver diseases. In the general population obesity is constantly and dramatically raising, and represents a global epidemics. In a study including both European and American patients, our group reported that in patients with compensated cirrhosis overweight/obesity is very frequently observed (55% OW, 15% OB in Spanish patients; > 50% OB in USA patients), being the figure similar to that of general population. Moreover, this study demonstrated that the increase in body mass index (BMI) is a risk factor for the development of decompensation of cirrhosis, independent of portal pressure and liver function (Berzigotti et al. Hepatology 2011). We also observed that included patients with cirrhosis and obesity showed a significant increase of portal pressure (estimated through hepatic venous pressure gradient measurement-HVPG), which was not found in OW or normal weight patients. This suggests that the mechanism inducing decompensation in obese patients with cirrhosis might be mediated by an increase in portal pressure, even if no data are available in this population to support this hypothesis. It is well known that in obesity the adipose tissue acquires a pro-inflammatory phenotype leading to increased release of IL-1, IL-6 and TNF-alfa and many other pro-fibrogenic cytokines and hormones, which might mediate also an increase in portal pressure.

Given these observation, and given the potential reversibility of OW/OB, we hypothesise that weight loss (obtained by diet and exercise) might effectively reduce the HVPG in patients with compensated cirrhosis and OW/OB, so reducing their risk to progression. We designed this proof-of-concept study to confirm this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years
* Compensated liver cirrhosis (diagnosed by biopsy or clear clinical, laboratory and imaging data), of any etiology; patients who presented decompensation due to gastroesophageal variceal hemorrhage can also be included if hemorrhage a) occurred > 3 months before inclusion AND b) has been treated with drugs+band ligation AND c) no other decompensations occurred simultaneously.
* HVPG > 5 mmHg
* BMI > 26 Kg/m2
* Absence of gastroesophageal varices or small esophageal varices OR large varices only if the patient is already on treatment with beta-blockers since at least 6 weeks.
* In case of presence of systemic arterial hypertension and/or diabetes, patients can be included if the treatment of these condition is stable for at least 3 months

Exclusion Criteria:

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
HVPG change | 4 months
  The effects of weight loss on portal pressure will be assessed by measuring the HVPG at baseline and after 4 months of diet+exercise in the included patients.

SECONDARY OUTCOMES:
Hepatic function | 4 months
  The effects of weight loss on liver function will be estimated by assessing standard liver tests and indocyanine green clearance at baseline and after 4 months of diet+exercise
Serum markers of fibrosis, angiogenesis, endothelial dysfunction and oxidative stress | 4 months
  The effects of weight loss on Serum markers of fibrosis, angiogenesis, endothelial dysfunction and oxidative stress will be assessed by extracting adequate blood samples at baseline and after 4 months of diet+exercise
Body adiposity changes | 4 months
  Changes in BMI and body fat% will be assessed by measuring body weight and % of fat at baseline and after 4 months of diet + exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Bosch, MD, Principal Investigator — Hospital Clinic and CIBERehd
Locations (6):
- Spain (6):
  - Hospital Clinic, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Vall D'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Universitario Ramón y Cajal, Madrid

REFERENCES:
- [Derived] Berzigotti A, Albillos A, Villanueva C, Genesca J, Ardevol A, Augustin S, Calleja JL, Banares R, Garcia-Pagan JC, Mesonero F, Bosch J; Ciberehd SportDiet Collaborative Group. Effects of an intensive lifestyle intervention program on portal hypertension in patients with cirrhosis and obesity: The SportDiet study. Hepatology. 2017 Apr;65(4):1293-1305. doi: 10.1002/hep.28992. Epub 2017 Mar 6. PMID 27997989